CLINICAL TRIAL: NCT04442516
Title: A Canadian Study of Cisplatin mEtabolomics and NephroToxicity
Brief Title: Cisplatin Induced Kidney Toxicity
Acronym: ACCENT
Status: Recruiting | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); London Health Sciences Centre (Other); Provincial Health Services Authority British Columbia (Other)
Responsible Party: Principal Investigator, Michael Zappitelli, Clinician Scientist, The Hospital for Sick Children
Other Study IDs: CisP Metabolomics
Record Dates: First submitted 2020-06-18; First posted 2020-06-22 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Acute Kidney Injury; Cancer
MeSH Terms: conditions — Acute Kidney Injury; Neoplasms | interventions — Surveys and Questionnaires; Urination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urinary and plasma metabolites and saliva or blood sample for DNA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adults receiving Cisplatin as part of their cancer therapy
  Interventions: Other: Questionnaire, sampling of blood, urine and saliva
- Children receiving Cisplatin as part of their cancer therapy
  Interventions: Other: Questionnaire, sampling of blood, urine and saliva

INTERVENTIONS:
Other: Questionnaire, sampling of blood, urine and saliva — We are following patients who are receiving Cisplatin as part of their cancer therapy.

SUMMARY:
Cisplatin (CisP) is a chemotherapeutic agent used to treat head and neck and lung cancer in adults and over 15 different pediatric cancers. Despite its known toxicity, CisP is still widely used as a first line chemotherapy as it is so effective. Nephrotoxicity is one of the most common adverse effects of CisP, occurring in 20-50% of patients. It manifests as acute kidney injury (AKI) typically within the first few days of exposure and is associated with short and long-term morbidity. Furthermore, AKI diagnosis is only possible once kidney damage has progressed to functional impairment, when mitigation strategies are ineffective. Tests that could predict AKI risk pre-emptively or diagnose early-stage AKI before functional loss would be very impactful, affording opportunities for prevention or early intervention to mitigate CisP nephrotoxicity, reduce morbidity and improve health outcomes.

The field of metabolomics seeks to identify patterns of small molecules (metabolites) involved in cell or tissue metabolism related to disease states, or patient factors like lifestyle and genetics. Plasma and urine are ideal for sampling the metabolome, which can identify at-risk patients and reveal disease-related changes earlier than existing diagnostic methods do.

In CisP-treated children and adults from across Canada, we will identify urine and plasma metabolite profiles a) prior to CisP dosing that predict CisP AKI risk, and b) shortly after dosing to identify early-stage nephrotoxicity, before clinical signs of AKI are detectable. Our identified biomarkers will allow individualization of CisP treatment based on the level of nephrotoxicity risk and the design of trials to mitigate the progression and complications of CisP nephrotoxicity.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants: Initiating treatment with CisP (≥75 mg/m2) for head/neck or lung cancers at one of the Adult participating sites; 18 years of age or older.
* Paediatric participants: Initiating treatment with CisP for any cancer diagnosis at one of the Pediatric participating sites; greater than 3 months of age.
* All participants: Consent to participate in the study.

Exclusion Criteria:

* Diagnosis of chronic kidney disease (CKD) at baseline (glomerular filtration rate <60 mL/min/1.73m2, determined by chart review of either formal glomerular filtration rate testing, 24 hour creatinine creatinine clearance of age-appropriate serum creatinine-based estimated glomerular filtration rate equations; past kidney transplant)
* Previous use of any nephrotoxic drugs included on the provided Excluded Nephrotoxic Medications list in the two weeks prior to initiation of CisP treatment
* Previous use of CisP
* Previous radiotherapy (total body irradiation or abdominal radiation only) in the last 1 month prior to study
* Previous hematopoietic stem cell transplant
* Any chronic or acute health condition that the investigator feels would render the patient inappropriate for this study, including but not limited to significant uncontrolled cardiorespiratory, hepatic, infectious, or renal disease at the discretion of the investigator

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Child Cohort. We already performed these study procedures on 159 children in the "ABLE" study, a 12-centre cohort study.Eligibility criteria and data/samples collected on these patients during their initial CisP treatment are almost identical to the present study. The cohort diagnoses include neuroblastoma, medulloblastoma, osteosarcoma, germ cell tumour, hepatoblastoma, and other cancers. Data and specimens from the pediatric study subjects in the ABLE study who were recruited during their first CisP infusion (about half) will be included in the current study. The remaining children (to reach a target of 300) will be recruited over 3 years from the following centres: McGill, UBC, SickKids, U. Manitoba and UWO. Adult Cohort. 300 adults (18 years of age or older) initiating CisP (≥75 mg/m2) treatment for head/neck or lung cancers will be recruited to participate in this study from PMH (Toronto), UBC and UWO over 2 years. Over 500 new patients/year are available across all sites.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-08-12 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
To identify patterns of metabolites and specific metabolites prior to and shortly after CisP treatment that predict AKI risk and identify the onset of AKI early (discovery cohort). | 8+ years

SECONDARY OUTCOMES:
To independently validate our findings and develop a precision medicine algorithm using metabolites to predict patients at high risk for developing CisP AKI (validation cohort). | 8+ years

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jain A, Huang R, Lee J, Jawa N, Lim YJ, Guron M, Abish S, Boutros PC, Brudno M, Carleton B, Cuvelier GDE, Gunaratnam L, Ho C, Adeli K, Kuruvilla S, Lajoie G, Liu G, Nathan PC, Rod Rassekh S, Rieder M, Waikar SS, Welch SA, Weir MA, Winquist E, Wishart DS, Zorzi AP, Blydt-Hansen T, Zappitelli M, Urquhart B. A Canadian Study of Cisplatin Metabolomics and Nephrotoxicity (ACCENT): A Clinical Research Protocol. Can J Kidney Health Dis. 2021 Nov 17;8:20543581211057708. doi: 10.1177/20543581211057708. eCollection 2021. PMID 34820133